CLINICAL TRIAL: NCT05778526
Title: Effectiveness of Social Virtual-reality on Enhancing Social Interaction Skills in Children With Attention-deficit/Hyperactivity Disorder: a Three-arm Pilot Randomised Controlled Trial
Brief Title: Social Virtual-reality on Enhancing Social Interaction Skills in Children With Attention-deficit/Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HSEARS20221221003
Record Dates: First submitted 2023-02-27; First posted 2023-03-21 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-06

CONDITIONS: Virtual Reality; Social Interaction; Attention-deficit/Hyperactivity Disorder
Keywords: Virtual reality; Social interaction; Attention-deficit/hyperactivity disorder; Three-arm pilot randomised controlled trial
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcomes assessor will be blinded to the study intervention period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social VR Intervention (Experimental): Social VR intervention is developed to enhance the social interaction skills of children. The participants will wear a head-mounted display for the Social VR intervention. Each session of the Social VR intervention lasts for a maximum of 20 minutes to ensure the participants focus on the intervention and prevent causing any physical effect. The duration will be adjusted depending on the emotion of the participants during the intervention. The Social VR intervention will mainly help the participant to enhance their social interaction skills and executive function. The intervention contains three real-life virtual scenarios, including (1) classroom and playground, (2) MTR station and compartment, and (3) supermarket and restaurant. One scenario will be adopted in each session. The sequences of the scenarios used in each session will be the same for all participants.
  Interventions: Behavioral: Virtual reality
- Traditional social skills training (Active Comparator): An experienced SEN teacher will teach the participants social interaction skills through tradidactic instructions and role-play activities. Four modules will be covered in the 3-week training: (1) how to introduce yourself and basic social skills; (2) how to listen to others; (3) how to share with others; (4) learn to know how people feel and how to empathise. These modules have been applied in many studies (Braswell & Bloomquist, 1991; Huang et al., 2015). The content of this training will be as similar as possible to the Social VR training. The training lasts 20 minutes which depends on the emotion of the participants.
  Interventions: Behavioral: Traditional social skills training
- Waitlist control group (No Intervention): The participants in this group will receive no training and they can participate in the social VR training after the intervention period. To ensure the consistency of the experiment, the participants are not allowed to initiate or change their pharmacological treatment during the 3-week intervention period.

INTERVENTIONS:
Behavioral: Virtual reality — There are a total of 12 training sessions for 3 weeks (4 sessions per week). Each session of the Social VR intervention lasts for a maximum of 20 minutes. The intervention contains three real-life virtual scenarios, including (1) a classroom and playground, (2) an MTR station and compartment, and (3) a supermarket and restaurant.
  Arms: Social VR Intervention
Behavioral: Traditional social skills training — There are a total of 12 training sessions for 3 weeks (4 sessions per week). Each session lasts for a maximum of 20 minutes. Four modules will be covered in the 3-week training: (1) how to introduce yourself and basic social skills; (2) how to listen to others; (3) how to share with others; (4) learn to know how people feel and how to empathise.
  Arms: Traditional social skills training

SUMMARY:
The study targets children with diagnosed ADHD and aims to (1) develop a social virtual reality-based intervention, (2) investigate its effects on improving the social skills and executive functioning of inhibitions, emotional control and attention of the children compared to traditional social skills training and (3) evaluate the subjects acceptability and compliance with social VR training for enhancing social interaction skills. It is hypothesised that the social interaction skills of the participants in the social VR training group are likely to perform better than those in the traditional social skills training group. Participants in the waitlist control group will receive no change in social interaction skills compared with the two intervention groups.

DETAILED DESCRIPTION:
The study will be a three-arm randomised controlled trial comparing the effects of social VR-based intervention with traditional social skills training on social skills and executive functioning of children with ADHD. Participants in the social VR intervention group and traditional social skill training group will receive 12 training sessions for 3 weeks (4 sessions per week), and participants in the waitlist control group will be asked to retain their usual lifestyles for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* aged between 6 and 12 years
* ethnic Chinese
* residing in Hong Kong
* having received a diagnosis of ADHD by Child Assessment Service in Hong Kong or via private practice
* stable on pharmacological and/or psychological treatment for ADHD 8 weeks before baseline (determined by health care professionals on the basis of medication data and behavioural observation)
* no initiation or change of pharmacological treatment for ADHD during the intervention period
* the ability to read Chinese, and speak and listen to Cantonese by the child and by at least one of their parents or legal guardian
* willing to provide informed consent by both participants and one of their parents or legal guardian

Exclusion Criteria:

* comorbid autism
* mental retardation
* an estimated IQ lower than 85 (using the Wechsler Intelligence Scale for Children - Fourth Edition (Hong Kong) (WISC-IV(HK)))
* autism spectrum disorder (previously diagnosed by health care professionals)
* comorbid acute psychiatric disorder (previously diagnosed by health care professionals)
* with a severe physical disability (e.g., blindness, deafness) or learning disability (e.g., dyslexia).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-02-18 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Qin, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- Ka Po WONG, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
It is confidential.

REFERENCES:
- [Derived] Wong KP, Zhang B, Lai CYY, Xie YJ, Li Y, Li C, Qin J. Empowering Social Growth Through Virtual Reality-Based Intervention for Children With Attention-Deficit/Hyperactivity Disorder: 3-Arm Randomized Controlled Trial. JMIR Serious Games. 2024 Oct 28;12:e58963. doi: 10.2196/58963. PMID 39467288
- [Derived] Wong KP, Qin J. Effectiveness of Social Virtual Reality Training in Enhancing Social Interaction Skills in Children With Attention-Deficit/Hyperactivity Disorder: Protocol for a Three-Arm Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Sep 18;12:e48208. doi: 10.2196/48208. PMID 37721790

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Social VR Intervention | Traditional Social Skills Training | Waitlist Control Group
Started | 30 | 30 | 30
Completed | 30 | 29 | 19
Not Completed | 0 | 1 | 11
Not completed — Lost to Follow-up | 0 | 1 | 3
Not completed — Protocol Violation | 0 | 0 | 8

BASELINE CHARACTERISTICS:
Population: (1) aged between 6 and 12 years; (2) Chinese ethnicity; (3) residing in Hong Kong; (4) having received a diagnosis of ADHD by Child Assessment Service in Hong Kong or via private practice; (5) stable on pharmacological and psychological treatment for ADHD 8 weeks before baseline; (6) no initiation or change of pharmacological treatment for ADHD during the intervention period; (7) ability to read Chinese and speak and listen to Cantonese by the child.
Groups:
- Total: Total of all reporting groups
Arm/Group | Social VR Intervention | Traditional Social Skills Training | Waitlist Control Group | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 30 | 90
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.63 (1.90) | 8.30 (1.70) | 8.67 (1.45) | 8.53 (1.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 6 | 17
  Male | 23 | 26 | 24 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 30 | 30 | 30 | 90
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 30 | 30 | 30 | 90
Having received a diagnosis of ADHD by Child Assessment Service in Hong Kong or via private practice [Count of Participants; unit: Participants] | 30 | 30 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Acceptability and Compliance
Description: The attendance of the participants during the trainings will be recorded. To verify the validity of the findings, training non-adherence of the participants will be terminated which will be stated in the consent form. The absence of any training session will be considered as non-adherence.
Time Frame: After 3 weeks
Measure: Number; unit: Percentage of sessions attended
Arm/Group | Social VR Intervention | Traditional Social Skills Training | Waitlist Control Group
Number analyzed (Participants) | 30 | 30 | 30
Percentage of sessions attended | 100 | 96.6 | 63.3

2. Secondary Outcome: Riggio Social Skills Inventory Assessment
Description: This assessment utilizes the Riggio Social Skills Inventory to objectively evaluate participants' social interaction skills. The total score ranges from 10 to 40, where higher scores indicate better social interaction skills. The inventory consists of 10 items, each scored on a scale from 1 (Never) to 4 (Always). Scores for each item are summed to compute a total score, with higher total scores representing better outcomes in social interaction skills. The inventory includes subscales that measure aspects of verbal and non-verbal communication.
Time Frame: 3 weeks post-intervention
Population: Data were collected from all participants who completed the assessments, including those from the waitlist control group who did not receive the intervention. This resulted in an analysis population of 30 participants in each group: 30 in the Social VR Intervention group, 30 in the Traditional Social Skills Training group, and 30 in the Waitlist Control group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social VR Intervention | Traditional Social Skills Training | Waitlist Control Group
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 38.20 (2.83) | 30.63 (6.57) | 24.50 (5.17)

3. Secondary Outcome: Social Skills Rating System - Parent Version (SSRS-P)
Description: This assessment evaluates participants' self-control, assertiveness, and initiative and cooperation. The SSRS-P consists of 3 subscales with a total of 31 items. A 3-point Likert scale (1 = Never, 2 = Sometimes, 3 = Often) is used for scoring. The total score ranges from 31 to 93, where higher scores indicate better social skills. Scores for each subscale are summed, contributing to the total score. The SSRS-P is a validated instrument commonly adopted in clinical trials of psychiatric and neurological disorders.
Time Frame: 3 weeks post-intervention
Population: Data were collected from the guardians of all participants who completed the SSRS-P assessments, resulting in 30 participants in each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social VR Intervention | Traditional Social Skills Training | Waitlist Control Group
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 33.33 (3.56) | 31.93 (2.78) | 31.50 (4.70)

4. Secondary Outcome: Behaviour Rating Inventory of Executive Function
Description: To assess the executive functioning of participants using the Behavior Rating Inventory of Executive Function (BRIEF), which will be scored by the participants' guardians. The subscales of inhibition (16 items) and emotional control (10 items) will be adopted in this study. A 3-point Likert scale (1 = Never, 2 = Sometimes, 3 = Often) is used to score. The total score ranges from 26 to 78, with higher scores indicating poor executive functions.
Time Frame: 3 weeks post-intervention
Population: Data were collected from the guardians of all participants who completed the BRIEF assessments, resulting in 30 participants in each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social VR Intervention | Traditional Social Skills Training | Waitlist Control Group
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 16.83 (3.08) | 17.98 (2.68) | 19.63 (4.91)

5. Secondary Outcome: Satisfaction of the Intervention
Description: Satisfaction with the intervention was measured using a 7-point Likert scale (1 = very dissatisfied, 7 = very satisfied) administered at the last session of the VR training group. The total score ranges from 1 to 7, with higher scores indicating greater satisfaction.
Time Frame: After the last session (after 3 weeks)
Population: Data were collected from 30 participants in the VR training group and 30 participants in the traditional social skills training group to assess satisfaction at the last session of the intervention.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Social VR Intervention | Traditional Social Skills Training
Number analyzed (Participants) | 30 | 30
Score on a scale | 6.8 (1.6) | 6.7 (1.7)

6. Secondary Outcome: Simulator Sickness Questionnaire
Description: To measure the motion sickness or physical discomfort of participants in VR environment. Nine items will be measured, including discomfort, fatigue, headache, eyestrain, sweating, nausea, difficulty concentrating, blurred vision and dizziness, with yes or no questions for each item.
Time Frame: Assessments will be conducted at the end of each session of the VR intervention group (twelve sessions in total), with the total score reflecting cumulative discomfort experienced across all sessions.
Population: Only the participants in the Social VR Intervention were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Social VR Intervention | Traditional Social Skills Training | Waitlist Control Group
Number analyzed (Participants) | 30 | 0 | 0
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline to 3 weeks post-intervention
Description: Standard adverse event definitions as per ClinicalTrials.gov were used for this study. Adverse events were systematically monitored throughout the intervention period. Participants were asked about any negative experiences at the beginning and end of each session, and researchers documented any observed adverse reactions during the sessions.
Arm/Group | Social VR Intervention | Traditional Social Skills Training | Waitlist Control Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT05778526/Prot_SAP_ICF_000.pdf